CLINICAL TRIAL: NCT00725777
Title: Efficacy and Safety of Artemether Lumefantrine Combination Therapy for the Treatment of Malaria Due to Plasmodium Ovale, Plasmodium Malariae, and Mixed Plasmodium Infections in Gabon
Brief Title: Treatment of Non-falciparum Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Schweitzer Hospital (Other)
Responsible Party: Principal Investigator, Michael Ramharter, Ass. Prof. PD, Albert Schweitzer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDC-08-01
Record Dates: First submitted 2008-07-14; First posted 2008-07-30 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Acute Non-falciparum Malaria
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: artemether-lumefantrine

INTERVENTIONS:
Drug: artemether-lumefantrine — Standard artemether-lumefantrine treatment

SUMMARY:
Patients with non-falciparum infection will be given artemether-lumefantrine for three days and will be followed up for 28 days. Besides efficacy and safety evaluations a substudy on immunology will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the age of 6 months and 60 years and with a minimum of 5kg bodyweight
* Presence of uncomplicated malaria confirmed by: i)fever or history of fever in the previous 4 days, and ii)positive microscopy of P. malariae or P. ovale or mixed infection with P.falciparum with parasite density > 50-200000/μl of blood
* Written informed consent

Exclusion Criteria:

* Patients with presence of other clinical conditions requiring hospitalization
* Presence of other febrile conditions
* Presence of significant anemia, defined by hemoglobin < 7g/dl
* Known history of hypersensitivity,allergic or adverse reactions to artemether or lumefantrine
* Intake of any antimalarial or antibiotics with known antimalarial activity in the preceding 2 weeks
* Pregnant and breast feeding females

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Parasitological cure rate on day 28 | D28

SECONDARY OUTCOMES:
Frequency and severity of drug related adverse events | D28

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Bélard, MD, Principal Investigator — Medical Research Unit of the Albert Schweitzer Hospital in Lambaréné
Locations (1):
- Medical Research Unit of the Albert Schweitzer Hospital, Lambaréné, Moyen-Ogooué Province, Gabon

REFERENCES:
- [Derived] Mombo-Ngoma G, Kleine C, Basra A, Wurbel H, Diop DA, Capan M, Adegnika AA, Kurth F, Mordmuller B, Joanny F, Kremsner PG, Ramharter M, Belard S. Prospective evaluation of artemether-lumefantrine for the treatment of non-falciparum and mixed-species malaria in Gabon. Malar J. 2012 Jul 10;11:120. doi: 10.1186/1475-2875-11-120. PMID 22515681